CLINICAL TRIAL: NCT04161313
Title: Comparison of Respiratory Function, Exercise Capacity and Peripheral Muscle Strength Among Patients With Cystic Fibrosis, Primary Ciliary Dyskinesia and Healthy Children
Brief Title: Respiratory Function, Exercise Capacity and Peripheral Muscle Strength Among Patients With CF, PCD and Healthy Children
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Lecturer in Department of Physiotheray and Rehabilitation, Bezmialem Vakif University
Other Study IDs: hdenizkulli2
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Primary Ciliary Dyskinesia; Cystic Fibrosis
Keywords: respiratory functions; exercise capacity; muscle strength
MeSH Terms: conditions — Ciliary Motility Disorders; Cystic Fibrosis | interventions — Respiratory Physiological Phenomena; Functional Residual Capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cystic fibrosis: children with cystic fibrosis
  Interventions: Other: Measurement of functional capacity; Other: pulmonary function test; Other: Functional capacity; Other: Peripheral muscle strength; Other: Respiratory muscle strength
- primary ciliary dyskinesia: children with primary ciliary dyskinesia
  Interventions: Other: Measurement of functional capacity; Other: pulmonary function test; Other: Functional capacity; Other: Peripheral muscle strength; Other: Respiratory muscle strength
- healthy controls: Age-matched healthy volunteers
  Interventions: Other: Measurement of functional capacity; Other: pulmonary function test; Other: Functional capacity; Other: Peripheral muscle strength; Other: Respiratory muscle strength

INTERVENTIONS:
Other: Measurement of functional capacity — Functional capacity of participants will be measured with six-minute walk test.
Other: pulmonary function test — It will be measured using basic spirometry and presented lung volume parameters such as FEV1,FVC,FEV1/FVC,PEF, FEF25-75
Other: Functional capacity — Functional capacity of participants will be measured with six-minute walk test and sit-to-stand test
Other: Peripheral muscle strength — Isometric M. Quadriceps strength will be measured using electronic hand held dynamometer in sitting position.
Other: Respiratory muscle strength — Inspiratory and expiratory muscle strength has been assessed by maximal inspiratory and expiratory mouth pressures.

SUMMARY:
The aim of this study is to compare pulmonary function, respiratory muscle strength, exercise capacity and peripheral muscle strength of patients with CF, PCD and healthy childrens.

DETAILED DESCRIPTION:
The impaired airway clearence and pulmonary functions, exercise intolerance, low physical activity level and decreased peripheral muscle strength make physiotherapy approaches important in the management of CF and PCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis or primary ciliary dyskinesia

Exclusion Criteria:

* Hospitalization history in past month
* Diagnosis of other chronic pediatric diseases which may impair exercise tolerance such as cerebral palsy or neuromuscular disease
* Candidates for lung transplantation or history of lung transplantation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with cystic fibrosis and primary ciliary dyskinesia and age matched healthy volunteers who do not have any diagnosed chronic diseases
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test distance | 15 minutes
  Distance walked in six minutes will be recorded in meters. Test will be conducted according to the guideline of American Thoracic Society (ATS).

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 5 minutes
  FVC will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Forced Expiratory Volume in 1 second (FEV1) | 5 minutes
  FEV1 will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Peak Expiratory Flow (PEF) | 5 minutes
  PEF will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
M. Quadriceps strength | 5 minutes
  Isometric M. Quadriceps strength (kg) will be measured using electronic hand held dynamometer in sitting position.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Denizoglu Kulli, PhD, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No